CLINICAL TRIAL: NCT04902131
Title: An Open-label, Randomised, 2-way Crossover, Single-dose, Bioequivalence Trial Comparing MENOPUR Solution for Injection in Pre-filled Pen and MENOPUR Powder and Solvent for Solution for Injection, After Subcutaneous Administration in Healthy Women
Brief Title: A Study Comparing MENOPUR in a Pen Formulation With a Powder and Solvent Formulation in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 000347
Record Dates: First submitted 2021-05-04; First posted 2021-05-26 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Injections; Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MENOPUR pen (Experimental)
  Interventions: Drug: A MENOPUR solution for injection in pre-filled pen, 600 IU/0.96 mL
- MENOPUR powder (Active Comparator)
  Interventions: Drug: A MENOPUR powder including solvent for solution for injection, 75 IU

INTERVENTIONS:
Drug: A MENOPUR solution for injection in pre-filled pen, 600 IU/0.96 mL — Single dose cross-over bioequivalence trial
  Other Names: Highly purified menotropin
  Arms: MENOPUR pen
Drug: A MENOPUR powder including solvent for solution for injection, 75 IU — Single dose cross-over bioequivalence trial
  Other Names: Highly purified menotropin
  Arms: MENOPUR powder

SUMMARY:
MENOPUR is a human menotrophin product, with a combination of human follicle-stimulating hormone (FSH) and luteinizing hormone (LH) activity. Human chorionic gonadotrophin (hCG) is the major contributor to the LH activity in the product. MENOPUR is approved in more than 130 countries for a variety of strengths and indications. In China, MENOPUR, 75 IU is approved for controlled ovarian hyperstimulation in relation to assisted reproductive technology (ART). The current trial is intended for supporting marketing authorization approval of a new formulation of MENOPUR in China.

MENOPUR is currently available in China as a powder and solvent for solution for injection, containing 75 IU of FSH and 75 IU of LH activity. A new liquid formulation is developed by Ferring Pharmaceuticals for administration with a disposable pre-filled injection pen, containing 600 IU of FSH and 600 IU of LH activity. MENOPUR solution for injection in pre-filled pen, 600 IU/0.96 mL is the test product and MENOPUR powder and solvent for solution for injection, 75 IU is the reference product in this trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Chinese women between the ages of 21 to 40 years at the time of signing the informed consent form
* Non-users or users of the combined oral contraceptive (COC) pill who describe experiencing menstrual cycles of 24 to 35 days in duration (both inclusive)
* Healthy according to medical history, physical and gynecological examinations, vital signs, 12-lead electrocardiogram, and laboratory tests in blood and urine
* Serum FSH levels ≤5 IU/L and estradiol levels ≤50 pg/mL on Day -3 and Day -1 in TP1

Key Exclusion Criteria:

* Any finding at the gynecological examination, transvaginal ultrasound or by cervical smear that is considered medically important
* A history of medical problems that could affect the functioning of the reproductive organs (ovaries and womb)
* A history of any medical problems that may prevent use of the combined hormonal contraceptive pill

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women, 21 to 40 years of age
Enrollment: 95 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of FSH: AUCt | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before investigational medicinal product [IMP] administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  AUCt is defined as area under the concentration-time curve from dosing to the last time point when the baseline adjusted concentration is above zero.
Pharmacokinetic parameter of FSH: Cmax | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  Cmax is defined as baseline adjusted maximum observed concentration.

SECONDARY OUTCOMES:
Pharmacokinetic parameter of FSH: AUCinf | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  AUCinf is defined as area under concentration-time curve from dosing to infinity using baseline adjusted concentrations.
Pharmacokinetic parameter of FSH: Tmax | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  Tmax is defined as time of maximum observed concentration.
Pharmacokinetic parameter of FSH: CL/F | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  CL/F is defined as apparent systemic clearance.
Pharmacokinetic parameter of FSH: Vz/F | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  Vz/F is defined as apparent volume of distribution during terminal phase.
Pharmacokinetic parameter of FSH: λz | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  λz is defined as first-order rate constant associated with the terminal (log-linear) portion of the concentration-time curve.
Pharmacokinetic parameter of FSH: t½ | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  t½ is defined as terminal half-life.
Pharmacokinetic parameter of human chorionic gonadotrophin (hCG): AUCt | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  AUCt is defined as area under the concentration-time curve from dosing to the last time point when the baseline adjusted concentration is above zero.
Pharmacokinetic parameter of hCG: AUCinf | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  AUCinf is defined as area under concentration-time curve from dosing to infinity using baseline adjusted concentrations.
Pharmacokinetic parameter of hCG: Cmax | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, 96, 120, 168 and 216 hours after administration
  Cmax is defined as baseline adjusted maximum observed concentration.
Pharmacokinetic parameter of LH: AUCt | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and 4, 8, 12, 24 and 48 hours after administration
  AUCt is defined as area under the concentration-time curve from dosing to the last time point when the baseline adjusted concentration is above zero.
Pharmacokinetic parameter of LH: Cmax | At -1, -0.5 hours pre-dose, and immediately pre-dose (within 10 min before IMP administration), and 4, 8, 12, 24 and 48 hours after administration
  Cmax is defined as baseline adjusted maximum observed concentration.
Frequency of adverse events (AEs) stratified by intensity | From signing of the informed consent up to the end-of-trial (11 to 18 days after the last IMP administration)
  The frequency of subjects with total AEs and AEs by categories of intensity (mild, moderate, severe) are presented.
  An AE was any untoward medical occurrence in a subject participating in clinical trial. The intensity of AE was classified using the following 3-point scale: mild = awareness of signs or symptoms, but no disruption of usual activities); moderate = disruption of usual activities (disturbing); or severe = inability to work or perform usual activities (unacceptable).
Frequency of injection site reactions stratified by intensity | Immediately after administration, and at 0.5 and 24 hours after administration on Day 1 and Day 2 of Treatment period 1 (TP1) and Time period 2 (TP2)
  The presence of injection site reactions (redness, pain, itching, swelling and bruising) immediately, 0.5 hours and 24 hours after the injection are presented.
  The injection site reactions were assessed as none, mild, moderate and severe. The number of injection site reactions (mild, moderate or severe) based on all assessments performed is presented.
Change from baseline of vital signs (systolic and diastolic blood pressure) | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Vital signs comprising systolic and diastolic blood pressure will be presented.
Change from baseline of vital sign (pulse) | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Vital sign comprising pulse will be presented.
Change from baseline of vital sign (body temperature) | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Vital sign comprising body temperature will be presented.
Change from baseline of 12-lead electrocardiogram (ECG): Heart rate | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (heart rate) parameter will be reported.
Change from baseline of 12-lead ECG: PR interval | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (PR interval) parameter will be reported.
Change from baseline of 12-lead ECG: RR interval | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (RR interval) parameter will be reported.
Change from baseline of 12-lead ECG: QRS interval | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (QRS interval) parameter will be reported.
Change from baseline of 12-lead ECG: QT interval | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (QT interval) parameter will be reported.
Change from baseline of 12-lead ECG: QTc interval | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (QTc interval) parameter will be reported.
Change from baseline of 12-lead ECG: QRS axis | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Change from baseline for 12-lead ECG (QRS axis) parameter will be reported.
Change from baseline of clinical chemistry: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameters including: Alanine aminotransferase, Alkaline phosphatase, Aspartate aminotransferase, and Gamma glutamyl transferase.
Change from baseline of clinical chemistry: Albumin | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Albumin.
Change from baseline of clinical chemistry: Glucose | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Glucose.
Change from baseline of clinical chemistry: Calcium | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Calcium.
Change from baseline of clinical chemistry: Chloride | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Chloride.
Change from baseline of clinical chemistry: Cholesterol | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Cholesterol.
Change from baseline of clinical chemistry: Phosphate | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Phosphate.
Change from baseline of clinical chemistry: Potassium | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Potassium.
Change from baseline of clinical chemistry: Sodium | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Sodium.
Change from baseline of clinical chemistry: Urea (blood urea nitrogen) | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Urea (blood urea nitrogen).
Change from baseline of clinical chemistry: C-reactive protein | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: C-reactive protein.
Change from baseline of clinical chemistry: Creatinine, Total bilirubin | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameters including: Creatinine, Total bilirubin.
Change from baseline of clinical chemistry: Thyroid stimulating hormone | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Thyroid stimulating hormone.
Change from baseline of clinical chemistry: Free triiodothyronine | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Free triiodothyronine.
Change from baseline of clinical chemistry: Free thyroxine | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Free thyroxine.
Change from baseline of clinical chemistry: FSH | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: FSH.
Change from baseline of clinical chemistry: Estradiol | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of clinical chemistry parameter including: Estradiol.
Change from baseline of haematology parameter: Haematocrit | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Haematocrit.
Change from baseline of haematology parameter: Haemoglobin | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Haemoglobin.
Change from baseline of haematology parameter: Mean cellular volume | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Mean cellular volume.
Change from baseline of haematology parameter: Mean corpuscular haemoglobin content | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Mean corpuscular haemoglobin content.
Change from baseline of haematology parameter: Mean corpuscular haemoglobin concentration | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Mean corpuscular haemoglobin concentration.
Change from baseline of haematology parameter: Red blood cell (RBC) count | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: RBC count.
Change from baseline of haematology parameter: Platelet count | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Platelet count.
Change from baseline of haematology parameter: Reticulocytes | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: Reticulocytes.
Change from baseline of haematology parameter: White blood cell count | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
  Blood samples were collected for the analysis of haematology parameter including: White blood cell count.
Change from baseline of urinalysis parameter: Protein | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Glucose | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Bilirubin | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: pH and Specific Gravity | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Nitrite | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Ketone | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Urobilinogen | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Blood | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)
Change from baseline of urinalysis parameter: Leukocytes | On Day -1 in TP1 and TP2, and at the follow-up (end-of-trial, 11 to 18 days after the last IMP administration) visit. Baseline is defined as pre-administration (Day -1)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (2):
- China (2):
  - Ferring investigational site, Nanjing, Gaoxin District
  - Ferring investigational site, Nanjing